CLINICAL TRIAL: NCT02431806
Title: A Double-blind, Placebo- and Active-Controlled Evaluation of the Safety and Efficacy of Levomilnacipran ER in Adolescent Patients With Major Depressive Disorder
Brief Title: Safety and Efficacy of Levomilnacipran ER in Adolescent Participants With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LVM-MD-11; NCT03087916 (obsolete NCT alias)
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Levomilnacipran; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received 2 dose matched over-encapsulated placebo capsules, once daily, orally during the Double-blind Treatment Period up to 8 weeks followed by a 1 week Taper-down Period if applicable as determined by the investigator.
  Interventions: Drug: Placebo
- Levomilnacipran 40 mg (Experimental): Participants received over-encapsulated levomilnacipran extended release (ER) 40 mg/day capsules orally starting at a dose of 10 mg/day on Day 1-2, 20 mg/day on Days 3-7 and 40 mg/day on Week 2 through Week 8 during the Double-Blind Treatment Period, followed by a 1-week Double-Blind Taper-down Period if applicable as determined by the investigator. Participants received 1 dose matched placebo capsule each day to maintain the blind.
  Interventions: Drug: Levomilnacipran
- Levomilnacipran 80 mg (Experimental): Participants received over-encapsulated levomilnacipran ER two 40 mg/day capsules (80 mg/day) orally starting at a dose of 10 mg/day on Day 1-2, 20 mg/day on Day 3-4, 40 mg/day on Day 5-7 and 80 mg/day on Week 2 through Week 8 during the Double-blind Treatment Period, followed by a 1-week Double-blind Taper-down Period if applicable as determined by the investigator. Participants received 1 dose matched placebo capsule the first week and during the taper-down period to maintain the blind.
  Interventions: Drug: Levomilnacipran
- Fluoxetine 20 mg (Active Comparator): Participants received over-encapsulated fluoxetine 20 mg/day tablets orally starting at a dose of 10 mg/day in Week 1 and 20 mg/day in Week 2 through Week 8 during the Double-blind Treatment Period, followed by a 1-week Double-blind Taper-down Period if applicable as determined by the investigator. Participants received 1 dose matched placebo capsule each day to maintain the blind.
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Placebo — Matched over-encapsulated placebo capsules administered orally on Day 1 to Week 8.
  Arms: Placebo
Drug: Levomilnacipran — Over-encapsulated levomilnacipran ER capsules administered orally on Day 1 to Week 8.
  Other Names: Fetzima
  Arms: Levomilnacipran 40 mg; Levomilnacipran 80 mg
Drug: Fluoxetine — Over-encapsulated fluoxetine tablets administered orally on Day 1 to Week 8.
  Other Names: Prozac
  Arms: Fluoxetine 20 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of levomilnacipran ER relative to placebo in adolescent outpatients (12-17 years) with Major Depressive Disorder (MDD). In addition, the study is designed to obtain pharmacokinetics (PK) data to guide dose selection for future pediatric studies of levomilnacipran.

DETAILED DESCRIPTION:
Study LVM-MD-11 is a randomized, double-blind, placebo- and active-controlled, parallel group, fixed-dose study in adolescent patients, ages 12-17 years. The study will be approximately 10 weeks in duration:

* 1-week screening/washout period
* 8-week double-blind treatment period
* 1-week double-blind down-taper period

Participants who meet the eligibility criteria at Visit 2 (Baseline) will be randomized to 1 of 4 treatment groups: placebo, levomilnacipran 40 mg/day, levomilnacipran 80 mg/day, or fluoxetine 20 mg/day.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female outpatients;12-17 years of age
* Meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for MDD, confirmed by Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children--Present and Lifetime (K-SADS-PL)
* Score ≥ 40 on the Children's Depression Rating Scale-Revised (CDRS-R) at Visits 1 and 2
* Clinical Global Impressions-Severity (CGI-S) score ≥ 4 at Visits 1 and 2
* Reliable caregiver
* Physical examination, vital signs, clinical laboratory tests, and electrocardiogram (ECG) normal or not clinically significant

Key Psychiatric Exclusion Criteria:

* DSM-IV-TR-based diagnosis of an axis I disorder other than MDD that is the primary focus of treatment
* Mental retardation or amnestic or other cognitive disorders
* Significant suicide risk:
* Suicide attempt within the past year OR
* Investigator judgment (based on psychiatric interview and Columbia-Suicide Severity Rating Scale (C-SSRS))

Key Treatment-Related Exclusion Criteria:

* Allergy, intolerance, or hypersensitivity to levomilnacipran, milnacipran, fluoxetine, or any other selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitors (SNRI)
* Use of prohibited concomitant medication that cannot be discontinued

Other Key Medical Exclusion Criteria:

* Any current medical condition that might interfere with the conduct of the study, confound the interpretation of study results, or affect participants safety
* Liver enzyme tests aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2X the upper limit of normal (ULN)
* Clinically significant cardiovascular disorders
* Seizure disorder or risk of seizure
* Drug or alcohol abuse or dependence (within the past year)
* Positive urine drug screen or blood alcohol

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 552 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Radecki, Study Director — Forest Research Institute, Inc., an affiliate of Allergan, plc
Locations (49):
- United States (48):
  - Harmonex, Inc, Dothan, Alabama
  - University of Arizona Department of Psychiatry, Tucson, Arizona
  - Advanced Research Center, Inc., Anaheim, California
  - ProScience Research Group, Culver City, California
  - Sun Valley Research Center, Imperial, California
  - Alliance for Research, Long Beach, California
  - Asclepes Research Centers, Panorama City, California
  - Syrentis Clinical Research, Santa Ana, California
  - Pacific Clinical Research Medical Group, Upland, California
  - MCB Clinical Research Center, Colorado Springs, Colorado
  - Florida Clinical Research Center; LLC, Bradenton, Florida
  - Coastal Clinical Research Specialists, Fernandina Beach, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Research in Miami Inc, Hialeah, Florida
  - Advanced Research Institute of Miami, Homestead, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - University of South Florida Board of Trustee, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Institute for Behavioral Medicine, Smyrna, Georgia
  - Clinical Research Institute, Stockbridge, Georgia
  - Sandeep Gaonkar, MD, Naperville, Illinois
  - NeuroMedical Institute, Panama, Illinois
  - Kentucky Pediatric Research, Bardstown, Kentucky
  - Adams Clinical Trials, LLC, Watertown, Massachusetts
  - Alivation Research, Lincoln, Nebraska
  - Kolade Research Institute, Las Vegas, Nevada
  - Healthy Perspectives - Innovative Mental Health Services. PLLC, Nashua, New Hampshire
  - Princeton Medical Institute, Princeton, New Jersey
  - Manhattan Behavioral Medicine, New York, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - Professional Psychiatric Services, Mason, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, Oklahoma City, Oklahoma
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - UTHSC-Houston, Houston, Texas
  - Bay Area Clinical Services dba Earle Research, Houston, Texas
  - Red Oak Psychiatry Associates, Houston, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
  - UVA Child and Family Psychiatry Clinic, Charlottesville, Virginia
  - Carilion Medical Center, Roanoke, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Eastside Therapeutic Resource dba Core Clinical, Everett, Washington
- INSPIRA Clinical Research, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Radecki DT, Robieson WZ, Gopalkrishnan M, Greenberg E, Aziz M. Safety and Efficacy of Levomilnacipran Extended Release in Pediatric Patients Aged 7-17 Years with Major Depressive Disorder: Results of Two Phase 3, Randomized, Double-Blind Studies. J Child Adolesc Psychopharmacol. 2024 Jun;34(5):241-250. doi: 10.1089/cap.2023.0080. Epub 2024 May 3. PMID 38700708

RESULTS

PARTICIPANT FLOW:
Groups:
- Levomilnacipran 40 mg/Day: Participants received over-encapsulated levomilnacipran extended release (ER) 40 mg/day capsules orally starting at a dose of 10 mg/day on Day 1-2, 20 mg/day on Days 3-7 and 40 mg/day on Week 2 through Week 8 during the Double-Blind Treatment Period, followed by a 1-week Double-Blind Taper-down Period if applicable as determined by the investigator. Participants received 1 dose matched placebo capsule each day to maintain the blind.
- Levomilnacipran 80 mg/Day: Participants received over-encapsulated levomilnacipran ER two 40 mg/day capsules (80 mg/day) orally starting at a dose of 10 mg/day on Day 1-2, 20 mg/day on Day 3-4, 40 mg/day on Day 5-7 and 80 mg/day on Week 2 through Week 8 during the Double-blind Treatment Period, followed by a 1-week Double-blind Taper-down Period if applicable as determined by the investigator. Participants received 1 dose matched placebo capsule the first week and during the taper-down period to maintain the blind.
- Fluoxetine 20 mg/Day: Participants received over-encapsulated fluoxetine 20 mg/day tablets orally starting at a dose of 10 mg/day in Week 1 and 20 mg/day in Week 2 through Week 8 during the Double-blind Treatment Period, followed by a 1-week Double-blind Taper-down Period if applicable as determined by the investigator. Participants received 1 dose matched placebo capsule each day to maintain the blind.
Period: Double-blind Treatment Period
Arm/Group | Placebo | Levomilnacipran 40 mg/Day | Levomilnacipran 80 mg/Day | Fluoxetine 20 mg/Day
Started | 142 | 136 | 139 | 135
Safety Population | 141 | 134 | 138 | 134
Completed | 117 | 115 | 107 | 109
Not Completed | 25 | 21 | 32 | 26
Not completed — Did not Receive Treatment | 1 | 2 | 1 | 1
Not completed — Adverse Event | 4 | 7 | 11 | 7
Not completed — Lack of Efficacy | 2 | 0 | 2 | 2
Not completed — Withdrawal of Consent | 10 | 7 | 5 | 5
Not completed — Lost to Follow-up | 7 | 4 | 5 | 8
Not completed — Investigational Product Non-compliance | 1 | 0 | 3 | 1
Not completed — Reason Not Specified | 0 | 1 | 5 | 2
Period: Double-blind Down-taper Period
Arm/Group | Placebo | Levomilnacipran 40 mg/Day | Levomilnacipran 80 mg/Day | Fluoxetine 20 mg/Day
Started | 111 | 109 | 104 | 107
Completed | 111 | 109 | 104 | 107
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants in the Randomized Population who took at least 1 dose of double-blind investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Levomilnacipran 40 mg/Day | Levomilnacipran 80 mg/Day | Fluoxetine 20 mg/Day | Total
Number analyzed (Participants) | 141 | 134 | 138 | 134 | 547
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (1.59) | 14.8 (1.62) | 14.8 (1.75) | 14.7 (1.67) | 14.7 (1.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 94 | 87 | 84 | 363
  Male | 43 | 40 | 51 | 50 | 184
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 36 | 32 | 36 | 137
  Not Hispanic or Latino | 108 | 98 | 106 | 98 | 410
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 1 | 3
  Asian | 1 | 1 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 52 | 46 | 49 | 40 | 187
  White | 81 | 81 | 83 | 88 | 333
  More than one race | 6 | 4 | 3 | 4 | 17
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Children's Depression Rating Scale-Revised (CDRS-R) Total Score [Mean (Full Range); unit: score on a scale] — CDRS-R is a 17-item scale measuring presence and severity of symptoms commonly associated with childhood depression and is scored on a 1-to-5- or 1-to-7-point scale. Rating of 1 indicates normal function. The CDRS-R total score ranges from 17 to 113; higher score indicates more severe depression. Population: Intent to Treat (ITT) Population included all participants in the Safety Population who had the baseline and at least 1 postbaseline assessment of the CDRS-R total score.
  score on a scale
    number analyzed (Participants) | 140 | 134 | 138 | 134 | 546
    (all) | 61.1 [40 to 83] | 61.8 [32 to 88] | 59.4 [41 to 81] | 61.5 [40 to 92] | 60.95 [32 to 92]
Clinical Global Impression-Severity (CGI-S) Scale [Mean (Full Range); unit: score on a scale] — The CGI-S is a clinician-rated scale used to rate the severity of the participant's current state of mental illness compared with major depressive disorder (MDD) population. The participant was rated on a scale from 1 to 7, where 1= Very much improved; 2= Much improved; 3= Minimally improved; 4= No change; 5= Minimally worse; 6= Much worse; 7= Very much worse. Higher score indicates worsening of mental illness. Population: ITT Population included all participants in the Safety Population who had the baseline and at least 1 postbaseline assessment of the CDRS-R total score. Overall number of participants analyzed is the number of participants with data available for analyses.
  score on a scale
    number analyzed (Participants) | 140 | 134 | 138 | 134 | 546
    (all) | 4.7 [4 to 6] | 4.8 [3 to 6] | 4.7 [4 to 6] | 4.7 [4 to 6] | 4.7 [3 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Children's Depression Rating Scale-Revised (CDRS-R) Total Score
Description: CDRS-R is a 17-item scale measuring presence and severity of symptoms commonly associated with childhood depression and is scored on a 1-to-5- or 1-to-7-point scale. Rating of 1 indicates normal function. The CDRS-R total score ranges from 17 to 113; higher score indicates more severe depression. A negative change from Baseline indicates improvement. Mixed Model for Repeated Measures (MMRM) was used for analysis.
Time Frame: Baseline (Week 0) to Week 8
Population: ITT Population included all participants in the Safety Population who had the baseline and at least 1 postbaseline assessment of the CDRS-R total score. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Levomilnacipran 40 mg/Day | Levomilnacipran 80 mg/Day | Fluoxetine 20 mg/Day
Number analyzed (Participants) | 118 | 115 | 110 | 112
score on a scale | -22.90 (1.09) | -23.28 (1.11) | -22.64 (1.12) | -24.37 (1.12)
Statistical Analysis 1: Comparison: Placebo vs Levomilnacipran 40 mg/Day; Test type: Superiority; p = 0.8035, Mixed Model Repeated Measures (MMRM); Least Squares (LS) Mean Difference = -0.38, 95% CI 2-sided [-3.41 to 2.64] — Estimates and p-values are based on MMRM with treatment group, pooled study center, visit, and treatment group-by-visit interaction as fixed effects, and baseline and baseline-by-visit as covariates using an unstructured covariance matrix
Statistical Analysis 2: Comparison: Placebo vs Levomilnacipran 80 mg/Day; Test type: Superiority; p = 0.8681, MMRM; LS Mean Difference = 0.26, 95% CI 2-sided [-2.80 to 3.31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Fluoxetine 20 mg/Day; Test type: Superiority; p = 0.3439, MMRM; LS Mean = -1.47, 95% CI 2-sided [-4.52 to 1.58] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Scale
Description: The CGI-S is a clinician-rated scale used to rate the severity of the participants current state of mental illness compared with MDD population. The participant was rated on a scale from 1 to 7, where 1= Very much improved; 2= Much improved; 3= Minimally improved; 4= No change; 5= Minimally worse; 6= Much worse; 7= Very much worse. Higher score indicates worsening of mental illness. A negative change from Baseline indicates improvement. MMRM was used for analysis.
Time Frame: Baseline (Week 0) to Week 8
Population: ITT Population included all participants in the Safety Population who had the baseline and at least 1 postbaseline assessment of the Children's Depression Rating Scale-Revised (CDRS-R) total score. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Levomilnacipran 40 mg/Day | Levomilnacipran 80 mg/Day | Fluoxetine 20 mg/Day
Number analyzed (Participants) | 118 | 115 | 110 | 112
score on a scale | -1.54 (0.10) | -1.52 (0.10) | -1.52 (0.10) | -1.68 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Levomilnacipran 40 mg/Day; Test type: Superiority; p = 0.8788, MMRM; LS Mean Difference = 0.02, 95% CI 2-sided [-0.25 to 0.29] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Levomilnacipran 80 mg/Day; Test type: Superiority; p = 0.9230, MMRM; LS Mean Difference = 0.01, 95% CI 2-sided [-0.26 to 0.29] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Fluoxetine 20 mg/Day; Test type: Superiority; p = 0.2895, MMRM; LS Mean Difference = -0.15, 95% CI 2-sided [-0.42 to 0.13] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: First dose of study treatment to end of study follow-up (Up to 10 Weeks)
Description: Safety Population included all participants in the Randomized Population who took at least 1 dose of double-blind investigational product.
Arm/Group | Placebo | Levomilnacipran 40 mg/Day | Levomilnacipran 80 mg/Day | Fluoxetine 20 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/134 | 0/138 | 0/134
Serious Adverse Events (participants affected / at risk) | 0/141 | 2/134 | 0/138 | 4/134
Other Adverse Events (participants affected / at risk) | 33/141 | 54/134 | 63/138 | 41/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=141) | Levomilnacipran 40 mg/Day (N=134) | Levomilnacipran 80 mg/Day (N=138) | Fluoxetine 20 mg/Day (N=134)
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=141) | Levomilnacipran 40 mg/Day (N=134) | Levomilnacipran 80 mg/Day (N=138) | Fluoxetine 20 mg/Day (N=134)
Tachycardia (Cardiac disorders) | 1 | 13 | 12 | 5
Nausea (Gastrointestinal disorders) | 8 | 19 | 22 | 5
Abdominal pain upper (Gastrointestinal disorders) | 4 | 6 | 7 | 4
Vomiting (Gastrointestinal disorders) | 3 | 11 | 11 | 4
Nasopharyngitis (Infections and infestations) | 3 | 4 | 7 | 7
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7 | 9 | 10
Headache (Nervous system disorders) | 15 | 20 | 19 | 13
Dizziness (Nervous system disorders) | 5 | 5 | 9 | 3
Somnolence (Nervous system disorders) | 3 | 6 | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT02431806/SAP_000.pdf
  • Study Protocol (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT02431806/Prot_001.pdf